CLINICAL TRIAL: NCT02111564
Title: Medically Ill Patient Assessment of Rivaroxaban Versus Placebo in Reducing Post-Discharge Venous Thrombo-Embolism Risk
Brief Title: A Study of Rivaroxaban (JNJ-39039039) on the Venous Thromboembolic Risk in Post-Hospital Discharge Patients
Acronym: MARINER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR103834; 2014-000305-13 (EudraCT Number); RIVAROXDVT3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-03-31; First posted 2014-04-11 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Respiratory Insufficiency; Stroke Acute; Infectious Diseases; Rheumatic Diseases
Keywords: Heart Failure; Respiratory Insufficiency; Stroke Acute; Infectious Diseases; Rheumatic Diseases; Medically ill Patient; Rivaroxaban; Thromboembolism; Prophylactic Anti-Coagulation
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency; Stroke; Communicable Diseases; Rheumatic Diseases; Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Each patient will receive either 10 mg or 7.5 mg rivaroxaban tablet once daily orally (by mouth) for 45 days. The dosing will depend on a creatinine clearance at screening.
  Interventions: Drug: Rivaroxaban, 10 mg; Drug: Rivaroxaban, 7.5 mg
- Placebo (Placebo Comparator): Each patient will receive matching placebo tablet once daily orally (by mouth) for 45 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban, 10 mg — Patients, randomly allocated to the rivaroxaban arm, with a creatinine clearance at screening greater than or equal to (>=)50 mL/min will receive 10 mg rivaroxaban tablet with or without food.
  Other Names: Xarelto; BAY59-7939
  Arms: Rivaroxaban
Drug: Rivaroxaban, 7.5 mg — Patients, randomly allocated to the rivaroxaban arm, with a creatinine clearance at screening from >=30 to less than (<)50 mL/min will receive 7.5 mg rivaroxaban tablet with or without food.
  Other Names: Xarelto; BAY59-7939
  Arms: Rivaroxaban
Drug: Placebo — All patients, randomly allocated to the placebo arm, will receive one placebo tablet with or without food.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rivaroxaban compared with placebo in the prevention of symptomatic venous thromboembolism (VTE) events and VTE-related death post-hospital discharge in high-risk, medically ill patients.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect)-controlled, event-driven, multicenter study in patients who are hospitalized for a specific acute medical illness and have other risk factors for venous thromboembolism (VTE). The study is designed to evaluate rivaroxaban in the prevention of symptomatic VTE events and VTE-related deaths for a period of 45 days post-hospital discharge. The study will consist of a screening phase, a 45-day double-blind treatment phase, and a 30-day follow-up phase. Study drug will start at randomization (Day 1), and will continue until Day 45 (inclusive). A total of approximately 12000 patients will be randomly assigned to either rivaroxaban or placebo in a 1:1 ratio. The total duration for a patient who completes the study after randomization is expected to be 75 days.

ELIGIBILITY:
Key Inclusion Criteria:

* The duration of the index hospitalization must have been at least 3 and no more than 10 consecutive days
* Must meet venous thromboembolism (VTE) risk criteria with a total modified Improve VTE Risk Score of: greater than or equal 4, or 3 with D-dimer > 2* upper limit of normal (ULN), or 2 with D-dimer > 2*ULN

Key Exclusion Criteria:

* Any serious bleeding within 3 months prior to randomization or occurring during index hospitalization
* Serious trauma (including head trauma) within 4 weeks before randomization
* History of hemorrhagic stroke at any time in the past
* Any medical condition that requires chronic use of any parenteral or oral anticoagulation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12024 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (595):
- United States (135):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Sheffield, Alabama
  - Scottsdale, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Fullerton, California
  - Los Angeles, California
  - Newport Beach, California
  - Orange, California
  - Sacramento, California
  - San Jose, California
  - San Marino, California
  - Santa Ana, California
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - Danbury, Connecticut
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Bay Pines, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Celebration, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Largo, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Saint Cloud, Florida
  - Sebring, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Wellington, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Normal, Illinois
  - North Chicago, Illinois
  - Hammond, Indiana
  - Lafayette, Indiana
  - Michigan City, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Topeka, Kansas
  - Alexandria, Louisiana
  - Lafayette, Louisiana
  - Metairie, Louisiana
  - Minden, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - Rockport, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Saginaw, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Bridgeton, Missouri
  - Columbia, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Atlantic City, New Jersey
  - Bridgewater, New Jersey
  - Marlton, New Jersey
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - Cortlandt Manor, New York
  - Jamaica, New York
  - Johnson City, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - New York, New York
  - Staten Island, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Maumee, Ohio
  - Springfield, Ohio
  - Willoughby, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Abington, Pennsylvania
  - Camp Hill, Pennsylvania
  - Chambersburg, Pennsylvania
  - Doylestown, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Johnstown, Pennsylvania
  - Lancaster, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Shippensburg, Pennsylvania
  - Pawtucket, Rhode Island
  - Columbia, South Carolina
  - Summerville, South Carolina
  - Athens, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Channelview, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Tyler, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Richland, Washington
  - Seattle, Washington
  - Huntington, West Virginia
  - La Crosse, Wisconsin
  - Marshfield, Wisconsin
- Argentina (15):
  - Bahía Blanca
  - Buenos Aires
  - Ciudad de Buenos Aires
  - Coronel Suárez
  - Corrientes
  - Córdoba
  - Esperanza
  - La Plata
  - Merlo
  - Morón
  - Munro
  - Rosario
  - San Miguel de Tucumán
  - Santa Fe
  - Santa Fé
- Australia (18):
  - Bedford Park
  - Box Hill
  - Caboolture
  - Cairns
  - Chermside
  - East Saint Kilda
  - Kogarah
  - Launceston
  - Lismore
  - Meadowbrook
  - Milton
  - Nedlands
  - Parkwood
  - Penrith
  - Redcliffe
  - South Brisbane
  - Sydney
  - VIC, Parkville
- Austria (5):
  - Feldkirch
  - Graz
  - Linz
  - Salzburg
  - Vienna
- Belarus (6):
  - Grodno
  - Homyel
  - Minsk
  - Mogilev
  - Vitebsk
  - Vychulki, Brest Region, Brest
- Bosnia and Herzegovina (7):
  - Banja Luka
  - Bihać
  - Foča
  - Mostar
  - Sarajevo
  - Tuzla
  - Zenica
- Brazil (18):
  - Belo Horizonte
  - Blumenau
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Canoas
  - Curitiba
  - Itajaí
  - Natal
  - Passo Fundo
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Salvador
  - Santo André
  - São José do Rio Preto
  - São Paulo
  - Votuporanga
- Bulgaria (18):
  - Blagoevgrad
  - Burgas
  - Dimitrovgrad
  - Gabrovo
  - Kozloduy
  - Lom
  - Lovech
  - Montana
  - Pernik
  - Pleven
  - Plovdiv
  - Razlog
  - Rousse
  - Sandanski
  - Sliven
  - Sofia
  - Veliko Tarnovo
  - Vidin
- Canada (13):
  - Edmonton, Alberta
  - Saint John, New Brunswick
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Jérôme, Quebec
  - Sherbrooke, Quebec
- Colombia (8):
  - Armenia
  - Barranquilla
  - Bogotá
  - Cali
  - Chía
  - Floridablanca
  - Medellín
  - Villavicencio
- Croatia (11):
  - Čakovec
  - Karlovac
  - Krapinske Toplice
  - Osijek
  - Pula
  - Rijeka
  - Šibenik
  - Virovitica
  - Zabok
  - Zadar
  - Zagreb
- Czechia (30):
  - Boskovice
  - Brno
  - Český Krumlov
  - Fryštát
  - Jablonec Na Nisou
  - Kladno
  - Krnov
  - Kyjov
  - Liberec
  - Litomyšl
  - Městec Králové
  - Nové Město na Moravě
  - Nymburk
  - Olomouc
  - Opava
  - Ostrava
  - Pardubice
  - Písek
  - Prague
  - Příbram
  - Slaný
  - Sternberk
  - Svitavy
  - Teplice
  - Trutnov
  - Třinec
  - Uherské Hradiště
  - Ústí nad Labem
  - Ústí nad Orlicí
  - Zlín
- Denmark (9):
  - Aalborg
  - Copenhagen
  - Esbjerg
  - Frederiksberg
  - Hellerup
  - Hilleroed
  - Hvidovre
  - København S
  - Roskilde
- Tallinn, Estonia
- Georgia (6):
  - Batumi
  - Kutaisi
  - Marneuli
  - Rustavi
  - Tbilisi
  - Telavi
- Germany (16):
  - Berlin
  - Coburg
  - Dresden
  - Esslingen am Neckar
  - Frankfurt
  - Heidelberg
  - Jülich
  - Karlsbad
  - Leipzig
  - Limburg
  - Mannheim
  - Minden
  - Mönchengladbach
  - Neuwied
  - Troisdorf
  - Witten
- Greece (11):
  - Achaïa
  - Alexandroupoli
  - Athens
  - Heraklion
  - Ioannina
  - Kifisia, Athens
  - Magoula
  - Pátrai
  - Thessaloniki
  - Thessalonikis
  - Voula
- Hungary (31):
  - Ajka
  - Baja
  - Balassagyarmat
  - Berettyóújfalú
  - Budapest
  - Cegléd
  - Debrecen
  - Eger
  - Farkasgyepü
  - Gödöllő
  - Gyõr
  - Gyula
  - Hódmezővásárhely
  - Kalocsa
  - Kaposvár
  - Kecskemét
  - Keszthely
  - Kistarcsa
  - Komárom
  - Miskolc
  - Nagykanizsa
  - Orosháza
  - Pécs
  - Sátoraljaújhely
  - Szeged
  - Szekszárd
  - Szentes
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Zalaegerszeg
- Israel (13):
  - Beersheba
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Modiin
  - Nahariya
  - Petah Tikva
  - Rehovot
  - Safed
  - Tel Litwinsky
  - Tiberias
- Latvia (9):
  - Balvi
  - Daugavpils
  - Jelgava
  - Jēkabpils
  - Krāslavas Apriņķis
  - Kuldīga
  - Liepāja
  - Riga
  - Ventspils
- Lithuania (8):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Tauragė
  - Utena
  - Vilniaus Apskritis
  - Vilnius
- Mexico (6):
  - Aguascalientes
  - Cuernavaca
  - Guadalajara
  - Mérida
  - Monterrey
  - San Pedro Garza García
- Netherlands (17):
  - 's-Hertogenbosch
  - Alkmaar
  - Almelo
  - Amsterdam
  - Arnhem
  - Harderwijk
  - Heerlen
  - Hoorn
  - Maastricht
  - Nieuwegein
  - Sittard-Geleen
  - Sneek
  - The Hague
  - Tilburg
  - Veldhoven
  - Zutphen
  - Zwolle
- North Macedonia (5):
  - Bitola
  - Ohrid
  - Shtip
  - Skopje
  - Struga
- Peru (2):
  - Callao
  - Lima
- Poland (30):
  - Bialystok
  - Bielsko-Biala
  - Bydgoszcz
  - Bystra
  - Czeladź
  - Gdynia
  - Kielce
  - Krakow
  - Kłodzko
  - Lodz
  - Lublin
  - Ostrołęka
  - Ostrów Mazowiecka
  - Oława
  - Pabianice
  - Poznan
  - Proszowice
  - Puławy
  - Płock
  - Rabka-Zdrój
  - Siedlce
  - Sopot,Gdynia
  - Sosnowiec
  - Szczecin
  - Tarn W N/a
  - Torun
  - Warsaw
  - Węgrów
  - Wroclaw
  - Łęczna
- Portugal (8):
  - Braga
  - Coimbra
  - Covilha
  - Figueira da Foz Municipality
  - Guimarães
  - Lisbon
  - Porto
  - Vila Nova de Gaia
- San Juan, Puerto Rico
- Romania (13):
  - Bacau
  - Baia Mare
  - Brasov
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Focşani
  - Iași
  - Oradea
  - Piteşti
  - Tg Mures
  - Timișoara
- Russia (21):
  - Arkhangelsk
  - Chelyabinsk
  - Irkutsk
  - Kazan'
  - Kemerovo
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Moskva
  - Novosibirsk
  - Orenburg
  - Penza
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tomsk
  - Ulyanovsk
  - Vsevolzhsk
  - Yaroslavl
  - Yekaterinburg
- Serbia (15):
  - Belgrade
  - Ćuprija
  - Čačak
  - Dedinje
  - Kamenitz
  - Kragujevac
  - Leskovac
  - Niš
  - Novi Sad
  - Smederevo
  - Subotica
  - Šabac
  - Valjevo
  - Vranje
  - Zaječar
- Slovakia (3):
  - Košice
  - Martin
  - Nitra
- South Africa (14):
  - Bellville
  - Bloemfontein
  - Cape Town
  - Durban
  - Durban Kwa Zulu Natal
  - Gatesville Cape Town
  - Groenkloof, Pretoria
  - Johannesburg
  - Kempton Park
  - Kuils River
  - Pretoria
  - Somerset West
  - Stellenbosch
  - Worcester
- Spain (39):
  - Alcalá de Henares
  - Alicante
  - Almería
  - Alzira
  - Aranjuez
  - Ávila
  - Balea
  - Barcelona
  - Burgos
  - Cartagena
  - Cáceres
  - Don Benito
  - Elche
  - Getafe
  - Granada
  - Huelva
  - Las Palmas de Gran Canaria
  - Logroño
  - Madrid
  - Majadahonda-Madrid
  - Málaga
  - Móstoles
  - Murcia
  - Olot
  - Oviedo
  - Palma de Mallorca
  - Pamplona
  - PAU de Sanchinarro
  - Sabadell
  - San Cristóbal de La Laguna
  - San Sebastián de los Reyes
  - Sant Boi de Llobregat
  - Sant Joan d'Alacant
  - Santander
  - Sarrià
  - Seville
  - Torrelavega Cantabria
  - Valencia
  - Zaragoza
- Turkey (Türkiye) (8):
  - Adana
  - Ankara
  - Antalya
  - Istanbul
  - Izmir
  - Konya
  - Rize
  - Samsun
- Ukraine (17):
  - Cherkasy
  - Chernihiv
  - Dnipropetrovsk
  - Ivano-Frankivsky
  - Kharkiv
  - Kherson
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (8):
  - Angus
  - Cardiff
  - Craigavon
  - Glasgow
  - Leeds
  - Manchester
  - Norwich
  - Plymouth

REFERENCES:
- [Background] Raskob GE, Spyropoulos AC, Zrubek J, Ageno W, Albers G, Elliott CG, Halperin J, Haskell L, Hiatt WR, Maynard GA, Peters G, Spiro T, Steg PG, Suh EY, Weitz JI. The MARINER trial of rivaroxaban after hospital discharge for medical patients at high risk of VTE. Design, rationale, and clinical implications. Thromb Haemost. 2016 Jun 2;115(6):1240-8. doi: 10.1160/TH15-09-0756. Epub 2016 Feb 4. PMID 26842902
- [Derived] Raskob GE, Ageno W, Albers G, Elliott CG, Halperin J, Maynard G, Steg PG, Weitz JI, Albanese J, Yuan Z, Levitan B, Lu W, Suh EY, Spiro T, Lipardi C, Barnathan ES, Spyropoulos AC. Benefit-Risk Assessment of Rivaroxaban for Extended Thromboprophylaxis After Hospitalization for Medical Illness. J Am Heart Assoc. 2022 Oct 18;11(20):e026229. doi: 10.1161/JAHA.122.026229. Epub 2022 Oct 7. PMID 36205248
- [Derived] Spyropoulos AC, Raskob GE, Cohen AT, Ageno W, Weitz JI, Spiro TE, Lu W, Lipardi C, Albers GW, Elliott CG, Halperin JL, Hiatt WR, Maynard G, Steg PG, Sugarmann C, Barnathan ES. Association of Bleeding Severity With Mortality in Extended Thromboprophylaxis of Medically Ill Patients in the MAGELLAN and MARINER Trials. Circulation. 2022 May 10;145(19):1471-1479. doi: 10.1161/CIRCULATIONAHA.121.057847. Epub 2022 Apr 7. PMID 35389229
- [Derived] Raskob GE, Spyropoulos AC, Spiro TE, Lu W, Yuan Z, Levitan B, Suh E, Barnathan ES. Benefit-Risk of Rivaroxaban for Extended Thromboprophylaxis After Hospitalization for Medical Illness: Pooled Analysis From MAGELLAN and MARINER. J Am Heart Assoc. 2021 Nov 16;10(22):e021579. doi: 10.1161/JAHA.121.021579. Epub 2021 Nov 10. PMID 34755519
- [Derived] Jamil A, Jamil U, Singh K, Khan F, Chi G. Extended Thromboprophylaxis With Betrixaban or Rivaroxaban for Acutely Ill Hospitalized Medical Patients: Meta-Analysis of Prespecified Subgroups. Crit Pathw Cardiol. 2021 Mar 1;20(1):16-24. doi: 10.1097/HPC.0000000000000232. PMID 32657973
- [Derived] Spyropoulos AC, Ageno W, Albers GW, Elliott CG, Halperin JL, Hiatt WR, Maynard GA, Steg PG, Weitz JI, Lu W, Spiro TE, Barnathan ES, Raskob GE. Post-Discharge Prophylaxis With Rivaroxaban Reduces Fatal and Major Thromboembolic Events in Medically Ill Patients. J Am Coll Cardiol. 2020 Jun 30;75(25):3140-3147. doi: 10.1016/j.jacc.2020.04.071. PMID 32586587
- [Derived] Weitz JI, Raskob GE, Spyropoulos AC, Spiro TE, De Sanctis Y, Xu J, Lu W, Suh E, Argenti D, Yang H, Albanese J, Lipardi C, Barnathan ES. Thromboprophylaxis with Rivaroxaban in Acutely Ill Medical Patients with Renal Impairment: Insights from the MAGELLAN and MARINER Trials. Thromb Haemost. 2020 Mar;120(3):515-524. doi: 10.1055/s-0039-1701009. Epub 2020 Jan 23. PMID 31975354
- [Derived] Spyropoulos AC, Ageno W, Albers GW, Elliott CG, Halperin JL, Hiatt WR, Maynard GA, Steg PG, Weitz JI, Suh E, Spiro TE, Barnathan ES, Raskob GE; MARINER Investigators. Rivaroxaban for Thromboprophylaxis after Hospitalization for Medical Illness. N Engl J Med. 2018 Sep 20;379(12):1118-1127. doi: 10.1056/NEJMoa1805090. Epub 2018 Aug 26. PMID 30145946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12024 participants were randomized (rivaroxaban-6007;placebo-6017). 5 participants in placebo were excluded(2 invalid consent,3 randomized before Health Authority approval).
Pre-assignment Details: Participants were randomized (1:1) to receive rivaroxaban or placebo. In rivaroxaban, participants were treated with rivaroxaban 10 mg or 7.5 mg as per their creatinine clearance level. Data in the participant flow section is reported for study discontinuation from the disposition data.
Groups:
- Rivaroxaban 10 mg or 7.5 mg: Participants with a creatinine clearance (CrCl) greater than or equal to (>=) 50 milliliter per minute (mL/min) received 10 milligram (mg) rivaroxaban tablet once daily orally and participants with a creatinine clearance from >=30 to less than (<) 50 mL/min at screening received 7.5 mg rivaroxaban tablet once daily orally for 45 days.
- Placebo: Participants received rivaroxaban matched placebo tablet once daily orally for 45 days.
Period: Overall Study
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Started | 6007 | 6012
Treated | 5982 | 5980
Completed | 5876 | 5869
Not Completed | 131 | 143
Not completed — Death | 109 | 120
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo | Total
Number analyzed (Participants) | 6007 | 6012 | 12019
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.06) | 69.7 (10.22) | 69.7 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2877 | 2858 | 5735
  Male | 3130 | 3154 | 6284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 499 | 482 | 981
  Not Hispanic or Latino | 5490 | 5510 | 11000
  Unknown or Not Reported | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 5 | 14
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 128 | 123 | 251
  Black or African American | 71 | 57 | 128
  White | 5782 | 5808 | 11590
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 120 | 122 | 242
  AUSTRALIA | 45 | 43 | 88
  AUSTRIA | 6 | 8 | 14
  BELARUS | 67 | 66 | 133
  BOSNIA-HERZEGOVINA | 298 | 299 | 597
  BRAZIL | 46 | 46 | 92
  BULGARIA | 714 | 714 | 1428
  CANADA | 21 | 22 | 43
  COLOMBIA | 70 | 70 | 140
  CROATIA | 135 | 135 | 270
  CZECH REPUBLIC | 115 | 116 | 231
  DENMARK | 3 | 4 | 7
  ESTONIA | 5 | 6 | 11
  GEORGIA | 880 | 882 | 1762
  GERMANY | 8 | 9 | 17
  GREECE | 66 | 65 | 131
  HUNGARY | 275 | 274 | 549
  ISRAEL | 55 | 56 | 111
  ITALY | 74 | 73 | 147
  LATVIA | 154 | 154 | 308
  LITHUANIA | 82 | 82 | 164
  MEXICO | 17 | 15 | 32
  NETHERLANDS | 8 | 9 | 17
  PERU | 33 | 32 | 65
  POLAND | 310 | 309 | 619
  PORTUGAL | 6 | 7 | 13
  PUERTO RICO | 0 | 1 | 1
  REPUBLIC OF MACEDONIA | 451 | 451 | 902
  ROMANIA | 162 | 162 | 324
  RUSSIAN FEDERATION | 571 | 571 | 1142
  SERBIA | 305 | 304 | 609
  SOUTH AFRICA | 103 | 102 | 205
  SPAIN | 192 | 191 | 383
  TURKEY | 35 | 35 | 70
  UKRAINE | 426 | 428 | 854
  UNITED KINGDOM | 4 | 4 | 8
  UNITED STATES | 145 | 145 | 290

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to First Occurrence of Composite of All Symptomatic Venous Thromboembolism (VTE) and VTE Related Death Adjudicated by Clinical Event Committee (CEC)
Description: Symptomatic VTE included lower extremity deep vein thrombosis (DVT) and non-fatal pulmonary embolism (PE). Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: Intention-to-treat (ITT) analysis set comprised all randomized participants who signed a valid informed consent, regardless of actual treatment received.
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 0.84 | 1.11
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.136, Cox proportional hazards model; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.52 to 1.09]

2. Primary Outcome: Event Rate Based on Time From Randomization to the First Occurrence of Major Bleeding Adjudicated by CEC
Description: A major bleeding event was defined using validated International Society on Thrombosis and Haemostasis (ISTH) bleeding criteria. A major bleeding event was defined as overt bleeding that was associated with a fall in hemoglobin of 2 gram per deciliter (g/dL) or more, or a transfusion of 2 or more units of packed red blood cells or whole blood, or a critical site defined as intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or a fatal outcome. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or last dose + 2 days.
Time Frame: From randomization to 2 days after the last dose (Day 45)
Population: The Safety analysis set included all enrolled participants in the ITT analysis set who received at least 1 dose of study drug.
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 5982 | 5980
Events per 100 participants in 45 days | 0.28 | 0.15
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.124, Cox proportional hazards model; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [0.84 to 4.23]

3. Secondary Outcome: Event Rate Based on Time From Randomization to First Occurrence of VTE-Related Death Adjudicated by CEC
Description: Event rate based on time from randomization to first occurrence of VTE-related death (adjudicated by CEC) was assessed. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: ITT analysis set comprised all randomized participants who signed a valid informed consent, regardless of actual treatment received.
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 0.72 | 0.77
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.751, Cox proportional hazards model; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.62 to 1.42]

4. Secondary Outcome: Event Rate Based on Time From Randomization to the First Occurrence of a Symptomatic Venous Thromboembolism Event (VTE) Adjudicated by CEC
Description: Event rate based on time from randomization to the first occurrence of a symptomatic VTE (adjudicated by CEC) was assessed. Symptomatic VTE included lower extremity DVT and non-fatal PE. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: as for outcome 3
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 0.19 | 0.42
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.023, Cox proportional hazards model; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.22 to 0.89]

5. Secondary Outcome: Event Rate Based on Time From Randomization to the First Occurrence of a Composite of Symptomatic VTE and All-Cause Mortality (ACM) Adjudicated by CEC
Description: Event rate based on time from randomization to the first occurrence of a composite of symptomatic VTE and ACM (adjudicated by CEC) was assessed. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: as for outcome 3
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 1.31 | 1.80
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.033, Cox proportional hazards model; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.54 to 0.97]

6. Secondary Outcome: Event Rate Based on Time From Randomization to the First Occurrence of a Composite of Symptomatic VTE, Myocardial Infarction (MI), Non-Hemorrhagic Stroke, and Cardiovascular (CV) Death Adjudicated by CEC
Description: Event rate based on time from randomization to the first occurrence of a composite of symptomatic VTE (lower extremity DVT and non-fatal PE), MI, non-hemorrhagic stroke, and CV death (death due to a known CV cause and death in which a CV cause cannot be ruled out; by this definition, a VTE-related death was considered a CV death) as adjudicated by CEC was reported. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: as for outcome 3
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 1.58 | 2.03
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.073, Cox proportional hazards model; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.60 to 1.02]

7. Secondary Outcome: Event Rate Based on Time From Randomization to First Occurrence of All-Cause Mortality (ACM) Adjudicated by CEC
Description: Event rate based on time from randomization to first occurrence of ACM (adjudicated by CEC) was assessed. Event rate was defined as number of events per 100 participants in 45 days of follow up. Participants who did not have events were censored on the minimum of last visit before or on death, or Day 45.
Time Frame: Up to Day 45
Population: as for outcome 3
Measure: Number; unit: Events per 100 participants in 45 days
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
Number analyzed (Participants) | 6007 | 6012
Events per 100 participants in 45 days | 1.19 | 1.49
Statistical Analysis 1: Comparison: Rivaroxaban 10 mg or 7.5 mg vs Placebo; Test type: Superiority; p = 0.156, Cox proportional hazards model; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.09]

ADVERSE EVENTS:
Time Frame: Up to 75 days (+/-5 days)
Description: Intention-to-treat (ITT) analysis set comprised all randomized participants who signed a valid informed consent, regardless of actual treatment received.
Arm/Group | Rivaroxaban 10 mg or 7.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 115/6007 | 126/6012
Serious Adverse Events (participants affected / at risk) | 475/6007 | 493/6012
Other Adverse Events (participants affected / at risk) | 250/6007 | 280/6012
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 mg or 7.5 mg (N=6007) | Placebo (N=6012)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute Left Ventricular Failure (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 3 | 1
Aortic Valve Incompetence (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 13 | 10
Atrial Flutter (Cardiac disorders) | 3 | 6
Atrioventricular Block Complete (Cardiac disorders) | 4 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 5 | 5
Cardiac Asthma (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 51 | 62
Cardiac Failure Acute (Cardiac disorders) | 14 | 14
Cardiac Failure Chronic (Cardiac disorders) | 13 | 8
Cardiac Failure Congestive (Cardiac disorders) | 24 | 25
Cardiac Valve Disease (Cardiac disorders) | 1 | 1
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 5 | 2
Cardiogenic Shock (Cardiac disorders) | 4 | 2
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiomyopathy Acute (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 4 | 4
Congestive Cardiomyopathy (Cardiac disorders) | 1 | 2
Cor Pulmonale (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Diastolic Dysfunction (Cardiac disorders) | 1 | 0
Hypertensive Heart Disease (Cardiac disorders) | 0 | 1
Interventricular Septum Rupture (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 1
Left Ventricular Failure (Cardiac disorders) | 4 | 2
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Fibrosis (Cardiac disorders) | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Nodal Rhythm (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Sinus Node Dysfunction (Cardiac disorders) | 2 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 2
Ventricular Tachycardia (Cardiac disorders) | 3 | 0
Motion Sickness (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Conjunctival Oedema (Eye disorders) | 1 | 0
Exophthalmos (Eye disorders) | 1 | 0
Retinal Artery Occlusion (Eye disorders) | 0 | 1
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Chronic Gastritis (Gastrointestinal disorders) | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 2
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1
Pancreatic Disorder (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 2 | 2
Peptic Ulcer (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Rectal Polyp (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 25 | 30
Fatigue (General disorders) | 1 | 2
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 2
Oedema Peripheral (General disorders) | 1 | 1
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 3
Sudden Cardiac Death (General disorders) | 1 | 2
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 3
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Hepatic Lesion (Hepatobiliary disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1
Breast Cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 5 | 3
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 11 | 10
Clostridium Difficile Colitis (Infections and infestations) | 2 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 1
Diabetic Foot Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 2
Endocarditis Bacterial (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1
Endotoxic Shock (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 3 | 4
Fungal Oesophagitis (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 3
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Haematoma Infection (Infections and infestations) | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Infectious Colitis (Infections and infestations) | 0 | 1
Infectious Pleural Effusion (Infections and infestations) | 1 | 0
Infective Exacerbation of Bronchiectasis (Infections and infestations) | 1 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 4
Infective Spondylitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Injection Site Abscess (Infections and infestations) | 1 | 0
Intervertebral Discitis (Infections and infestations) | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 58 | 48
Pneumonia Bacterial (Infections and infestations) | 2 | 4
Pneumonia Pseudomonal (Infections and infestations) | 0 | 1
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 0 | 2
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis Chronic (Infections and infestations) | 2 | 1
Pyoderma (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 3 | 3
Sepsis (Infections and infestations) | 4 | 3
Septic Shock (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1
Splenic Abscess (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 2 | 0
Systemic Infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0
Tuberculous Pleurisy (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 11 | 11
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 4
Viral Infection (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 3
Head Injury (Injury, poisoning and procedural complications) | 1 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Intestinal Anastomosis Complication (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1
Nerve Injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 1
Twiddler's Syndrome (Injury, poisoning and procedural complications) | 0 | 1
Aspiration Bronchial (Investigations) | 1 | 0
Body Temperature Increased (Investigations) | 0 | 2
Cardiac Output Decreased (Investigations) | 1 | 0
Myocardial Necrosis Marker Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Vertebral Lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Infiltration Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Malignant Neoplasm of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mediastinum Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Craniocervical Syndrome (Nervous system disorders) | 1 | 0
Demyelinating Polyneuropathy (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Facial Paralysis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0
Hypoglycaemic Encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1
Orthostatic Intolerance (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 5
Vascular Encephalopathy (Nervous system disorders) | 0 | 1
Vertebral Artery Stenosis (Nervous system disorders) | 1 | 0
Vertigo CNS Origin (Nervous system disorders) | 1 | 0
Device Dislocation (Product Issues) | 0 | 1
Device Failure (Product Issues) | 1 | 0
Device Occlusion (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Conversion Disorder (Psychiatric disorders) | 0 | 1
Panic Attack (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 7 | 8
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 2
Ketonuria (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 2 | 0
Renal Failure (Renal and urinary disorders) | 3 | 3
Renal Impairment (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 3 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 81 | 77
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lupus Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary Pneumatocele (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Vasculitic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Bereavement (Social circumstances) | 0 | 1
Immobile (Social circumstances) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Aortic Dissection (Vascular disorders) | 0 | 1
Aortic Stenosis (Vascular disorders) | 2 | 1
Arterial Stenosis (Vascular disorders) | 1 | 0
Distributive Shock (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypertensive Crisis (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 5 | 3
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Artery Occlusion (Vascular disorders) | 1 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 0 | 2
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Post Thrombotic Syndrome (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 mg or 7.5 mg (N=6007) | Placebo (N=6012)
Diarrhoea (Gastrointestinal disorders) | 69 | 52
Headache (Nervous system disorders) | 114 | 147
Hypertension (Vascular disorders) | 75 | 93

LIMITATIONS AND CAVEATS:
Study was stopped prior to achieving preplanned 161 participants with primary outcome events. Other limitations included how VTE-related death was defined and participants with moderate renal impairment may have been under-dosed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT02111564/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT02111564/SAP_001.pdf